CLINICAL TRIAL: NCT03944993
Title: Effects of Pulsed Electromagnetic Fields (PEMFS) On Cerebral Haemodynamics - EPOCH Study
Brief Title: Effects of Pulsed Electromagnetic Fields (PEMFS) On Cerebral Haemodynamics
Acronym: EPOCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Premature termination due to logistical limitations.
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPOCH1.0
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2019-05

CONDITIONS: Cerebral Hemodynamics; Cognitive Change
Keywords: PEMF; Prefrontal cortex; Exercise mimetic; Pulsed Electromagnetic Fields

STUDY DESIGN:
Intervention Model Description: The study is designed as a double-blinded, randomised, controlled pilot study. As a pilot study, 33 healthy adults will be enrolled and randomised into the intervention or sham arm at 2:1 ratio. Within the intervention arm, 50% of the participants will receive PEMFs in the non-dominant leg and the remaining 50% will receive intervention in the dominant leg (n = 11, 11). There are no restrictions based on race or gender.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulsed Electromagnetic Field Therapy (Dominant leg) (Experimental): Active Pulsed Electromagnetic Field therapy; exposed once weekly for 10 minutes on dominant leg.
  Interventions: Device: Pulsed Electromagnetic Fields Therapy (Dominant leg)
- Pulsed Electromagnetic Field Therapy (Non-dominant leg) (Experimental): Active Pulsed Electromagnetic Field therapy; exposed once weekly for 10 minutes on non-dominant leg.
  Interventions: Device: Pulsed Electromagnetic Fields Therapy (Non-dominant leg)
- Sham Therapy (Control) (Sham Comparator): Inactive Pulsed Electromagnetic Field therapy; exposed once weekly for 10 minutes.
  Interventions: Device: Sham Therapy (Control)

INTERVENTIONS:
Device: Pulsed Electromagnetic Fields Therapy (Dominant leg) — Participants of this arm will be exposed to 10 minutes of Pulsed Electromagnetic Fields on their dominant leg once a week for a total of 6 weeks. A minimum of 5-day and maximum of 9-day interval between each treatment session shall be followed.
  The PEMF device produces pulsed magnetic fields at flux densities up to 1.5 mT peak.
  Other Names: PEMF; MRegen
  Arms: Pulsed Electromagnetic Field Therapy (Dominant leg)
Device: Pulsed Electromagnetic Fields Therapy (Non-dominant leg) — Participants of this arm will be exposed to 10 minutes of Pulsed Electromagnetic Fields on their non-dominant leg once a week for a total of 6 weeks. A minimum of 5-day and maximum of 9-day interval between each treatment session shall be followed.
  The PEMF device produces pulsed magnetic fields at flux densities up to 1.5 mT peak.
  Other Names: PEMF; MRegen
  Arms: Pulsed Electromagnetic Field Therapy (Non-dominant leg)
Device: Sham Therapy (Control) — Participants of this arm will be not be exposed to the fields. Sham treatment will utilise the same PEMF apparatus for 10 minutes, but in non-operational mode, which is indistinguishable from when the apparatus is in operation. Duration of intervention is 6 weeks. A minimum of 5-day and maximum of 9-day interval between each treatment session shall be followed.
  Arms: Sham Therapy (Control)

SUMMARY:
The investigators are looking to determine the effects of PEMFs device on cerebral blood flow and cognition in healthy volunteers. Through in vitro tests and in vivo animal studies, the investigators have shown that at an extremely low flux density (strength) of 1 millitesla (mT) and with short exposures of 10 minutes a week, PEMFs can recapitulate many of the healthful benefits of exercise without imparting a mechanical stress on the tissues and cells.

In the first-in-man study, 10 healthy volunteers were exposed to PEMFs for 6 weeks with 10 minutes of field exposure per week, and experienced an average increase of 30% in leg strength. No side effects were reported.

In this study, the investigators aim to understand the cerebral effects of an exercise mimetic (PEMFs) via the muscle milieu.

DETAILED DESCRIPTION:
Human and animal studies have reported the beneficial influence of exercise on cognitive and brain functions. Accordingly, exercise is drawing increasing research attention as a possible lifestyle factor for improving neurocognitive functions.

Low frequency and low amplitude Pulsed Electromagnetic Fields (PEMFs) recapitulate many of the benefits of exercise by activating many of the same cellular second messenger cascades activated by mechanical input (exercise) yet, without imparting a physical stress on the cells. Through a series of in vitro and in vivo experiments the investigators have shown that at field strengths of 1-2 mT amplitude, the PEMF system stimulates muscle without physically stressing the tissues and delivers the following benefits: 1) slows muscle loss, 2) improves muscle strength and, 3) releases important regenerative and metabolism-enhancing agents.

Functional near-infrared spectroscopy (fNIRS) is a relatively new optical imaging technology that uses light in the near-infrared spectrum to non-invasively monitor the haemodynamic responses evoked by neural activity through measuring the changes in oxyhaemoglobin (HbO) and deoxyhaemoglobin (HbR) concentrations in the cerebral cortex. The increased blood supply to the area of neural activation typically results in an increase in HbO concentration while a decrease is observed in HbR due to the blood's washout effect. The HbO and HbR responses from fNIRS measurements have been shown to be spatially and temporally correlated with the blood oxygen level-dependent signal obtained by fMRI. The advantage of fNIRS over other imaging modalities is that it is inexpensive, non-invasive, non-ionising and portable, making it a highly popular modality for implementing brain-computer interfaces. OBELAB NIRSIT is a commercially available, high-density fNIRS device that optically measures haemodynamic variations in the pre-frontal cortex (PFC).

Low-frequency and low amplitude pulsed electromagnetic fields (PEMFs) recapitulate many of the healthful benefits of exercise by activating many of the same cellular second messenger cascades activated by mechanical input (exercise) yet, without imparting a physical stress on the cells. Response windows are a largely unrecognised rule in mechanobiological systems, whereby cells are most responsive to a given strain, duration and frequency of stimulation; greater strain of higher frequency and duration of stimulation is too much of a stress for cells and results in null responses.

The investigators have shown that PEMFs likewise obey an electromagnetic window of efficacy with temporal and frequency dependencies of similar scale as those required for mechanical stimulation, further supporting the conclusion that PEMFs are activating cellular mechanotransduction pathways. At field strengths of 1-2 mT amplitude, the PEMF system stimulates muscle without physically stressing the tissues and aims to deliver the following benefits: 1) slows muscle loss; 2) improves muscle strength and; 3) releases important regenerative and metabolism-enhancing agents. Accordingly, this study will investigate the exercise mimetic effects of PEMFs on cerebral haemodynamics and cognitive performance via targeting muscle. The results of this study will support future work with patients with memory deficits, such as mild cognitive impairment, to possibly mitigate disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21- 65 years
* Ability to provide informed consent

Exclusion Criteria:

* Received any investigational drug or device within 30 days prior to study baseline visit or is enrolled in another clinical trial
* History of cardiac, neurological, or rheumatic diseases
* History of malignancy within the past 5 years
* Undergone surgery of any type within the past 6 months
* Anticipated need for surgery of any type during the next 3 months
* Previous treatment with the study device
* Metal implants in the lower limb
* Existing or planned pregnancy
* Lactating women
* Leg circumference > 63 cm
* Colour vision deficiency

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Change in cerebral haemodynamic responses | Baseline and Week 7
  The frontal lobe activity of the participants will be measured pre- and post-PEMF stimulation. We will then use the modified Beer-Lambert law (MBLL) to extract haemodynamics data from that signal after applying filtering to reject noise. Haemodynamics data of the three treatment groups will be incorporated into regression analysis. The amplitude of the signal will be further normalised by dividing the averaged values by the standard deviation during the first 10 seconds before task onset. The coordinates of the head landmarks and probe positions will be used to estimate the centroid position of each channel in the Montreal Neurological Institute standard brain space. We will calculate the Area Under Curve (AUC) of the waveform of averages and normalised HbO and HbR during the task. The AUC values of the fNIRS signals between pre- and post-PEMF stimulation in the PFC will be compared by paired t-tests to confirm changes.
Change in cognitive performance | Baseline and Week 7
  To determine any cognitive improvement as a result of PEMF from baseline using Stroop task.

SECONDARY OUTCOMES:
Quadriceps muscle strength | Baseline and Week 7
  To determine the extent leg dominancy affects PEMF response in muscles i.e. percentage increase in quadriceps strength compared to baseline.
Thigh girth | Baseline and Week 7
  To determine the extent leg dominancy affects PEMF response in muscle, we will measure participants' thigh girth (cm) 5 cm above from the superior border of the patella.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Franco-Obregon, Principal Investigator — National University of Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parate D, Franco-Obregon A, Frohlich J, Beyer C, Abbas AA, Kamarul T, Hui JHP, Yang Z. Enhancement of mesenchymal stem cell chondrogenesis with short-term low intensity pulsed electromagnetic fields. Sci Rep. 2017 Aug 25;7(1):9421. doi: 10.1038/s41598-017-09892-w. PMID 28842627
- [Background] Crocetti S, Beyer C, Schade G, Egli M, Frohlich J, Franco-Obregon A. Low intensity and frequency pulsed electromagnetic fields selectively impair breast cancer cell viability. PLoS One. 2013 Sep 11;8(9):e72944. doi: 10.1371/journal.pone.0072944. eCollection 2013. PMID 24039828
- See also: News article covering MRegen — https://www.straitstimes.com/singapore/health/nus-team-creates-magnetic-device-to-aid-muscle-recovery